CLINICAL TRIAL: NCT01549860
Title: IN-BALANCE VLU Inflammation, Bacteria, & Angiogenesis Effects in Launching Venous Leg Ulcer Healing
Brief Title: Effects of Non Contact Low Frequency Ultrasound in Healing Venous Leg Ulcers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Celleration, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IN-BALANCE VLU
Record Dates: First submitted 2012-03-07; First posted 2012-03-09 (Estimated); Results first posted 2015-07-30 (Estimated); Last update posted 2015-07-30 (Estimated); Status verified 2015-07

CONDITIONS: Venous Insufficiency; Venous Reflux; Lower Extremity Ulcer
Keywords: Venous Insufficiency; Reflux; Lower Extremity Ulcer
MeSH Terms: conditions — Venous Insufficiency; Leg Ulcer; Gastroesophageal Reflux

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Standard of Care (No Intervention): 30 to 40 mmHg compression, dressing for moist wound healing environment, debridement as needed. Minimum of one treatment per week and up to 3 times per week per investigator discretion for 4 weeks
- SOC + Mist Therapy (Experimental): 30 to 40 mmHg compression, dressing for moist wound healing environment, debridement as needed plus non-contract low frequency ultrasound 3 x per week for 4 weeks.
  Interventions: Device: MIST Therapy

INTERVENTIONS:
Device: MIST Therapy — Non-contact low frequency ultrasound therapy
  Arms: SOC + Mist Therapy

SUMMARY:
This trial is a prospective, randomized, controlled, multi-center study of subjects presenting with chronic lower extremity venous ulcers. The study will evaluate the safety and effectiveness of MIST Therapy® plus standard of care (MIST+SOC) compared to Standard of Care (SOC) alone in the treatment of lower extremity venous ulcers.

DETAILED DESCRIPTION:
The study compared the treatment effect of non-contact low frequency ultrasound in addition to standard of care versus standard of care alone in healing chronic venous leg ulcers in subjects who had documented venous stasis and reflux. Subjects that were screened and met the major inclusion criteria received standardized treatment of 30 to 40 mmHg compression, moist wound healing dressings, and debridement for a two week run-in period. If their study ulcer did not decreased by greater than 30% they were eligible for randomization. The primary endpoint was wound area reduction after four (4) weeks of study treatment. The study was performed at 22 study centers. The study included two sub-studies: fluid and tissue analysis and a wound recidivism registry that are ongoing.

ELIGIBILITY:
Inclusion Criteria:

* Lower extremity full thickness venous ulcer of > 30 days duration
* Subject's wound must be between 4 cm² and 50 cm² at screening
* Documented ABI that is between 0.8 and 1.2 on the study limb or transcutaneous partial pressure oxygen (TcpO2) > 40 mmHG; or a toe pressure > 40 mmHG; or a Doppler waveform consistent with adequate flow in the foot (biphasic or triphasic waveforms) at time of screening
* Biopsy for wounds > 6 months duration
* Documented index wound etiology of venous stasis with reflux and /or incompetent valves

Exclusion Criteria:

* Index ulcer wound that is less than 1 cm in distance from another ulcer wound
* > 5 ulcers on the index leg
* Index ulcer wound has exposed tendons, ligaments, muscle, or bone
* Index ulcer wound presents with clinical signs of acute infection, suspected or known
* Subjects with evidence of osteomyelitis or cellulitis or gangrene in the study limb
* Subjects with amputation above a Trans Metatarsal Amputation (TMA) in the study limb
* Subjects with active malignancy on the study limb except non-melanoma skin cancer
* Index ulcer that is of arterial disease etiology
* Index ulcer of other primary etiology (ie. vasculitis, arterial, pyoderma)
* Subjects with planned vascular surgery, angioplasty or thrombolysis procedures within the study treatment phase
* Subjects with planned surgical procedure during the study treatment phase for the index wound including skin flap or skin graft
* Subjects within 6 weeks postoperatively of a vascular o skin graft procedure.
* Subject has had prior skin replacement, negative pressure therapy, or traditional ultrasound therapy applied to the index wound in the 14 days prior to screening
* Subject has had ultrasound treatment (including MIST Therapy) of the index wound.
* Subject has received growth factor therapy (e.g., autologous platelet-rich plasma gel, becaplermin, bilayered cell therapy, dermal substitute, extracellular matrix) within 14 days of screening date.
* Subject is currently receiving or has received radiation or chemotherapy within 3 months of randomization.
* Female subjects that are pregnant or refuse to utilize adequate contraceptive methods and are of childbearing age during the trial.
* Subject has one or more medical condition(s), uncontrolled diabetes (i.e. HbA1c > 12), renal, hepatic, hematologic, neurologic, or immune disease that in the opinion of the investigator would make the subject an inappropriate study candidate
* Subject's wound would require ultrasound near an electronic implant or prosthesis
* Subject is known to be suffering from a disorder or other situation that the subject or investigator feels would interfere with compliance or other study requirements
* Subject is currently enrolled or has been enrolled in the last 30 days in another investigational device or drug trial

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 156 (Actual)
Dates: Start 2012-04; Primary Completion 2014-05 (Actual); Study Completion 2015-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gary Gibbons, MD, Principal Investigator — South Shore Hospital; Vicki Driver, DPM, Principal Investigator — Providence RI
Locations (1):
- South Shore Hospital, Weymouth, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 156 subjects were consented for the study, 112 subjects met the major inclusion/exclusion criteria (study cohort), 81 subject were randomized (reduced <30% during run-in period).
Groups:
- Standard Care (SC): 30 to 40 mmHg compression, dressing for moist wound healing environment, debridement as needed. Minimum of one treatment per week and up to 3 times per week per investigator discretion for 4 weeks
- SC + Mist Therapy: 30 to 40 mmHg compression, dressing for moist wound healing environment, debridement as needed plus non-contract low frequency ultrasound 3 x per week for 4 weeks.
  MIST Therapy: Non-contact low frequency ultrasound therapy
Period: Overall Study
Arm/Group | Standard Care (SC) | SC + Mist Therapy
Started | 40 | 41
Completed | 38 | 40
Not Completed | 2 | 1
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Physician Decision | 1 | 1

BASELINE CHARACTERISTICS:
Population: Eligible subjects randomized
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard Care (SC) | SC + Mist Therapy | Total
Number analyzed (Participants) | 40 | 41 | 81
Age, Continuous [Median (Full Range); unit: years] | 60.0 [34.0 to 81.0] | 58.0 [33.0 to 86.0] | 59.0 [33.0 to 86.0]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 13 | 24
  Male | 29 | 28 | 57
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 11 | 13 | 24
  White | 24 | 22 | 46
  More than one race | 5 | 6 | 11
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 40 | 41 | 81
BMI [Median (Full Range); unit: kg per meter squared] | 33.2 [21.2 to 55.7] | 37.4 [17.2 to 69.7] | 34.7 [17.2 to 69.7]
Wound Age at Randomization [Median (Full Range); unit: months] | 8.9 [1.7 to 204.5] | 10.3 [1.5 to 114.0] | 10.3 [1.5 to 204.5]
Wound Area at Randomization [Median (Full Range); unit: centimeters squared] | 9.8 [2.5 to 36.9] | 12.4 [3.1 to 53.3] | 11.0 [2.5 to 53.3]

OUTCOME MEASURES:

1. Primary Outcome: Wound Area Mean Percent Reduction
Description: Compare between the treatment groups percent wound area reduction at four weeks of study treatment.
  H0: µMIST+SC -- µSC = 0 HA: µMIST+SC -- µSC ≠ 0 Where µ = percent reduction in wound size.
Time Frame: 4 weeks post baseline visit (randomization visit)
Population: eligible subjects that were randomized
Measure: Mean (Standard Deviation); unit: percentage of mean area reduction
Arm/Group | Standard Care (SC) | SC + Mist Therapy
Number analyzed (Participants) | 40 | 41
percentage of mean area reduction | 45.8 (32.5) | 61.6 (28.9)
Statistical Analysis 1: Comparison: Standard Care (SC) vs SC + Mist Therapy; Test type: Superiority or Other; p < 0.024, t-test, 2 sided

2. Secondary Outcome: Heal Rates
Description: Compare rate of wound closure between study arms for 12 weeks post randomization. Descriptive statistics as not a powered endpoint.
Time Frame: 12 weeks post randomization
Population: Eligible subjects randomized
Measure: Number; unit: participants
Arm/Group | Standard Care (SC) | SC + Mist Therapy
Number analyzed (Participants) | 40 | 41
participants | 10 | 16

3. Secondary Outcome: Change in Pain VAS Scores
Description: Compare VAS Pain Scores between arms at baseline and 4 weeks post randomization
  Subjects indicate their pain level by drawing a mark on a 10 cm line on a visual analog scale (VAS) at randomization and 4 week post treatment visit. The left end of the line indicates "no pain" and the right end of line indicates "worst pain imaginable". VAS score is determined by using a ruler placed at 0 (left end of scale) and measuring the distance from zero to the patient's mark . The objective is to compare the change in VAS values in MIST+SC to SC alone.
  H0: The average change in pain level is not different between MIST and SC HA: The average change in pain level is different between MIST and SC H0: µMIST = µSC vs HA: µMIST ≠ µSC,
  Statistical Analysis. A repeated measures ANCOVA will be used to test for differences in change in VAS with an indicator variable to indicate treatment, any demographic variables which were significant in the baseline comparisons.
Time Frame: Baseline, 2 weeks and 4 weeks post randomization
Population: Eligible Subjects Randomized
Measure: Median (Full Range); unit: VAS pain level measured in centimeters
Arm/Group | Standard Care (SC) | SC + Mist Therapy
Number analyzed (Participants) | 40 | 41
VAS pain level measured in centimeters
  Randomization (baseline) VAS Score | 3.0 [0.0 to 9.0] | 3.0 [0.0 to 10.0]
  4 Week post-randomizaton VAS Score | 2.4 [0.0 to 10.0] | 0.6 [0.0 to 9.1]
Statistical Analysis 1: Comparison: Standard Care (SC) vs SC + Mist Therapy; Test type: Superiority or Other; p < 0.0126, ANCOVA — The MIST+SOC subjects decreased in their reported mean pain scores and reduced from a median of 3.0 to 0.6 cm after four weeks of study treatment

ADVERSE EVENTS:
Time Frame: Throughout 12 week study
Description: Only device or study procedure related adverse events were collected in this post market study
Arm/Group | Standard Care (SC) | SC + Mist Therapy
Serious Adverse Events (participants affected / at risk) | 0/40 | 0/41
Other Adverse Events (participants affected / at risk) | 0/40 | 0/41

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No